## **INFORMED CONSENT FORM**

## Psychological Monitoring of Victims of Terrorism and Effectiveness of Psychological Treatments

(October 10th, 2011)

## RESEARCH PROJECT ON PSYCHOLOGICAL MONITORING OF VICTIMS OF TERRORISM AND EFFECTIVENESS OF PSYCHOLOGICAL TREATMENTS

## DECLARATION OF VOLUNTARY PARTICIPATION

Through this document I consent to voluntarily participate in this study on the psychological follow-up of victims of terrorism and the effectiveness of psychological treatments.

I understand that I will be conducting several interviews and will be asked to complete several questionnaires asking about my physical and mental health, about my thoughts, behaviors and feelings, and about the terrorist attack(s) I have suffered, and about other events that have affected me. I understand that my responses will be completely confidential, that I may not answer any questions I do not wish to answer, and that I may refuse to complete any questionnaire, interview, or instrument and withdraw from the research at any time without prejudice to myself.

I also understand that I give my consent to voluntarily participate in a psychological treatment program for victims of terrorist attacks in order to try to improve my health and well-being and reduce the negative psychological consequences produced by the terrorist attack(s) that I have suffered. This psychological treatment program involves:

- 1. Weekly attendance at therapeutic sessions on the date and time established by the therapists during the duration of the program.
- 2. Perform those therapeutic tasks that are entrusted to me, which will be specifically aimed at improving my health and well-being.

I have been informed that I can leave the treatment program at any time without prejudice to myself and that the interviewer will answer any of my questions for the purposes of this study, however, certain questions that may affect the results will not be answered until completion.

I have been informed and I understand that the study does not intend to collect information on specific people, and that all data will be coded while maintaining my anonymity. I consent that the results of this study may be published in scientific journals or books or disseminated by other means to the scientific community. However, I understand that my name will never appear in said media, that the writings will only reflect the group results and that the identity of the participants will be protected.

I have been informed that any question that concerns me about any aspect of this study can be raised directly with Dr. María Paz García Vera, Full Professor of the Department of Clinical Psychology at the Complutense University of Madrid and Director of this study (phone: 913942614; e-mail: <a href="mailto:mpgvera@psi.ucm.es">mpgvera@psi.ucm.es</a>).

I have read and I understand the explanations abovementioned, and I agree to participate in this study.

Signed:

Participant Signature:
Signed:\_\_\_\_\_\_
Investigator Statement

The undersigned, researcher of the study "Psychological follow-up of victims of terrorism", has presented this information to the participant, has asked him about any question that may have arisen in this regard, has answered their questions to the best of his/her knowledge and has obtained their consent.

Researcher's signature: